CLINICAL TRIAL: NCT06786858
Title: Home Training for Upper Limb Stroke Rehabilitation Using a Hand Exoskeleton
Brief Title: Hand Exoskeleton Training Study
Acronym: HandMATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00004431
Record Dates: First submitted 2023-03-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- HandMate Use (Experimental): HandMate device fitted for a stroke participant.
  Interventions: Device: HandMate

INTERVENTIONS:
Device: HandMate — HandMate device is used for 20 hours in 4 weeks. Device is then used in the home for 3 months at discretion of participant.

SUMMARY:
The goal of this study is to evaluate the HandMATE device's effectiveness in the rehabilitation of stroke patients and asses if the HandMATE application is received well by stroke survivors.

Participants will use the HandMate device in clinic and in the home. They will also complete clinical upper extremity assessments.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of novel device and its potential to help stroke victims regain functional use of their hand and regain independent living. The study will also evaluate the potential of the device to be used at home, this would allow increased therapy intensity and decreased overall treatment costs (fewer therapist hours required and decreased travel costs).

ELIGIBILITY:
Inclusion Criteria:

* Age of 21 or older
* diagnosis of stroke more than 6 months prior confirmed from MRI or CT
* voluntary hand activity (score of 1 or more, finger extension item, Fugl-Meyer Test)
* adequate cognitive status
* Impaired ability to open affected hand

Exclusion Criteria:

* hemispatial neglect
* severe sensory loss (2 or more on the sensory item, NIH Stroke Scale/Score)
* receiving or planning to receive antispasticity medications during enrollment into the study
* less than full passive range of motion in finger joints
* receiving physical or occupational therapy outside of study protocols
* have excessive pain in any joint of the affected extremity that could limit ability to cooperate with the protocols

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity (FMA-UE) Test | Change from baseline Fugl-Meyer score at 6 weeks
  Evaluates and measures recovery in post-stroke hemiplegic patients. The FMA-UE Test will assess upper limb motor impairments for this study. It is a 33-item test that measures motor and reflex function in the upper body. Each item is scored on a scale of 0-2, with 0 indicating inability, 1 indicating beginning ability, and 2 indicating normal. The total score ranges from 0-66, highest score indicating no disability.
Action Research Arm Test (ARAT) | Change from baseline ARAT score at 6 weeks
  The ARAT is 19-item clinical assessment used to measure the functional ability of the upper extremity, particularly in individuals recovering from a stroke, by evaluating their performance on tasks like grasping, gripping, pinching, and gross arm movements. It is scored on a four-level ordinal scale (0-3). Highest score indicating normal movement.
Motor Activity Log | Change from baseline MAL score at 6 weeks
  The Motor Activity Log will be used to assess use of the limb at home. Respondents rate how they use their more-impaired arm for activities of daily living (ADLs) in the home (brushing teeth, buttoning a shirt, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Pete Lum, PhD, Principal Investigator — MedStar RI
Locations (1):
- MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States